CLINICAL TRIAL: NCT02832687
Title: A Multi-center, Randomized, Double-blind, Pilot Study on the Effect of Intravenous Multi-dose Acetaminophen on Readiness for Discharge in Patients Undergoing Surgery With General Anesthesia
Brief Title: Multi-dose Acetaminophen for Patients Undergoing General Anesthesia
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was halted due to the worldwide COVID-19 pandemic and the cancellation of all elective cases.
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Principal Investigator, Michal Gajewski, Assistant Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 20150002613
Record Dates: First submitted 2016-05-24; First posted 2016-07-14 (Estimated); Results first posted 2021-12-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: Recovery Following Cholecystectomy
MeSH Terms: interventions — Acetaminophen; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- normal saline (Active Comparator): Patients will receive 100 milliliters of normal saline with the first dose given preoperatively in the holding area followed by re-dosing every four hours from that point up to a maximum of 4 doses in 24 hours. Blinded medication will be prepared by research pharmacist.
  Interventions: Drug: normal saline
- acetaminophen (Experimental): Patients 50kg or more will receive either 1000mg IV acetaminophen with the first dose given preoperatively in the holding area followed by re-dosing every four hours from that point up to a maximum of 4 doses or 4000mg in 24 hours. Patients <50 kg will receive 12.5mg/kg to a maximum of 75 mg /per kg/per day as per the label dose with repeat dosing Q4 hours. Blinded medication will be prepared by research pharmacist in 100mL of normal saline
  Interventions: Drug: Acetaminophen

INTERVENTIONS:
Drug: Acetaminophen — patients 50kg or more receive1000mg in 100milliliters of normal saline every 4 hours to a maximum dose 4000mg/24 hours. <50kg receive 12.5mg/kg to a maximum of 75mg/kg/24 hours.
  Other Names: Ofirmev
  Arms: acetaminophen
Drug: normal saline — 100mL of normal saline every 4 hours to a maximum administration of 400mL
  Other Names: placebo
  Arms: normal saline

SUMMARY:
Study Objective The aim of the proposed study is to examine the effect of Q4 hour multidose IV acetaminophen on patients' readiness for discharge. In doing so the investigators will also investigate the various factors that could potentially contribute to a patient's readiness for discharge such as overall opioid consumption, time to rescue medication, incidence of postoperative nausea and vomiting, pain scores, and perioperative stress markers and their overall correlation with IV acetaminophen intake.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, two-arm parallel study.. Patients 50kg or more will receive either 1000mg IV acetaminophen or placebo with the first dose given preoperatively in the holding area followed by re-dosing every four hours from that point up to a maximum of 4 doses or 4000mg in 24 hours. Patients <50 kg will receive 12.5mg/kg to a maximum of 75 mg /per kg/per day as per the label dose with repeat dosing Q4 hours.

After pre-oxygenation, general anesthesia will be induced with lidocaine (1 mg/kg Ideal Body Weight), propofol (1-2 mg/kg Actual Body Weight), and fentanyl (up to 5 mcg/kg Actual Body Weight). Additionally all subjects with receive 2 mg midazolam. Tracheal intubation will be facilitated with rocuronium (0.6 - 1.2 mg/kg Actual Body Weight). Anesthesia will be maintained with air/oxygen (60%/40%) and desflurane. A remifentanyl infusion (0.05-2mcg/kg/min Ideal Body Weight) will be continued throughout the entire case with no further analgesics being administered. All patients will receive ondansetron 4 mg prior to the end of operation as well as additional antiemetics in the PACU as judged by the attending anesthesiologist. Patients will be awakened and extubated in the OR meeting standard extubation criteria. Once extubated all patients will then be transferred to the PACU where they will be assessed via the SPEEDs criteria 5 minutes after arrival and then every 15 minutes for the duration of their PACU stay. While in the PACU, all patients will be assessed for pain using the Visual Analog Scale. Pain will be treated as per our protocol with 0.2mg IV hydromorphone for mild pain (VAS 1-3), 0.4 mg IV hydromorphone for moderate pain (VAS 4-6), and 0.6 mg IV hydromorphone (VAS 7-10). As soon as a patient meets all the SPEEDs criteria he/she will be transferred to phase II of the recovery. In phase II, if need be, pain will be managed according to the following orders: 0.2mg intravenous hydromorphone for mild pain (VAS 1-3), 0.4 mg intravenous hydromorphone for moderate pain (VAS 4-6) and 0.6mg intravenous hydromorphone for severe pain (VAS 7-10).

The patient's readiness for discharge will be our primary outcome. Each patient will be assessed within 5 minutes of arriving in the PACU and then every 15 minutes thereafter until subject reaches maximum score. The assessment will be done using the SPEEDs criteria, which has recently been shown to be as specific and more sensitive for phase 1 nursing interventions and therefore more accurate in predicting which patients are fast-track eligible as compared to the standard Modified Aldrete 2 and Fast-Track criteria (38).

The secondary outcomes will include:

1. Post-operative pain scores a. Assessed every 15 minutes during the recovery period using the Visual and Numerical Analog Scales for 2 hours and then every 4 hours thereafter until discharge.
2. Time to first rescue medication a. 0.2mg intravenous hydromorphone for mild pain (VAS 1-3) b. 0.4mg intravenous hydromorphone for moderate pain (VAS 4-6) c. 0.6 mg intravenous hydromorphone for severe pain (VAS 7-10)
3. Total dosage of post-operative opioids given.
4. Incidence of post operative nausea and vomiting and need for additional antiemetics.
5. Phase II satisfaction survey:

a. This will focus on three of the following factors rated on a scale of 1 to 5, with 1 being dissatisfied/unlikely while 5 being most satisfied/very likely.

i. How satisfied are you with the overall experience? ii. How likely are you to recommend this anesthetic and analgesic to others? iii. How likely would you ask for a similar anesthetic and analgesic in the future if need be? f) Concentration of the plasma stress markers including cortisol, norepinephrine, epinephrine, and C Reactive Protein (CRP).

a. Changes in mediator levels in the IV acetaminophen versus placebo groups will be compared. Plasma samples will be collected before administration of any drug (after placement of IV lines), before incision, and 60 minutes after arrival in PACU. Blood [15millLiters] will be collected at the time points described above from an additional intravenous catheter placed in the patient's arm. These specimens will be placed in vacutainer tubes with no anti-coagulant. Blood will be drawn with a syringe attached directly to the angiocatheter which has been placed intravenously. To prevent hemolysis, blood will be transferred without a needle, to a vacutainer whose top has been removed. The vacutainer top will be replaced and specimens labeled with study name, subject's study IDentification number, sample number (1, 2, 3,), and dated. Bloods from the first two time points will be kept refrigerated until the final sample is obtained postoperatively. They will be centrifuged, serum removed, aliquoted and stored at -80 degrees C until analysis. All samples will be run in duplicate on with plates and reagents of the same lot. Any samples varying greater than 15% between duplicates

ELIGIBILITY:
Inclusion Criteria:

* Undergoing ambulatory laparoscopic cholecystectomy.
* American Society of Anesthesiologists physical status 1, 2 or 3.-

Exclusion Criteria -

* Cognitively impaired (by history) and unable or unwilling to consent
* Chronic steroid or opioid user (as prescribed for a chronic systemic illness)
* Parturient or nursing mother. Patients who have been informed by a physician that they have liver or kidney disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2017-06-19 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michal Gajewski, Do, Principal Investigator — Rutgers, State University of New Jersey
Locations (3):
- United States (3):
  - New Jersey Medical School, Newark, New Jersey
  - University Hospital, Newark, New Jersey
  - New York Methodist Hospital, Brooklyn, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Planned enrollment was "90" whereas the actual enrollment was "88".
Pre-assignment Details: At the time when recruitment reached 88 subject, elective surgeries at our institution were paused because of pandemic. However, when elective surgeries were resumed, Mallinckrodt, Inc. who provided support for the study filed for bankruptcy and we were not longer able to continue recruitment.
Period: Overall Study
Arm/Group | Normal Saline | Acetaminophen
Started | 41 | 47
Participants Who Were Included in the Analysis | 31 | 34
Completed | 41 | 45
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 2

BASELINE CHARACTERISTICS:
Population: A total of 88 patients were enrolled; from 47 who were randomized to receive intravenous acetaminophen 45 completed the study; from 41 received placebo 41 completed. A total of 65 patients were included into analyses with 34 receiving intravenous acetaminophen and 31 receiving placebo.
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Saline | Acetaminophen | Total
Number analyzed (Participants) | 31 | 34 | 65
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Median (q1, q3)
  years | 40 [28 to 56] | 44 [33 to 59] | 42 [31 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 25 | 51
  Male | 5 | 9 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 5 | 11 | 16
  White | 3 | 4 | 7
  Hispanic | 23 | 19 | 42
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 31 | 34 | 65
ASA Physical Status [Count of Participants; unit: Participants]
  The American Society of Anesthesiologists (ASA) Physical Status I (Patient is healthy) | 12 | 6 | 18
  ASA Physical Status II (Patient has mild systemic disease) | 18 | 26 | 44
  ASA Physical Status III (Patient has severe systemic disease that is not incapacitating) | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Readiness for Discharge
Description: Number (percentage) of Participants with Readiness for Discharge (achieving discharge-readiness status at end of 2- hours post-surgery evaluated using the SPEEDs criteria: oxygen saturation, pain control, emesis control, extremity movement, dialogue, and stable vital signs.
Time Frame: 2 hours following surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Saline | Acetaminophen
Number analyzed (Participants) | 31 | 34
Participants | 26 | 33

2. Secondary Outcome: Post Operative Pain Scores
Description: Pain scores every 15 min for 2 hours or until achieving discharge-readiness, whatever comes first, an average of 1 hour.
  Visual Analogue Scale (VAS) for pain was used: score on a scale from 0 (no pain) to 10 (worst pain) were recorded.
Time Frame: Every 15 min for 2 hours or until achieving discharge-readiness, whatever comes first, an average of 1 hour
Population: Not all participants were analyzed at every time point up to 120 minutes but only until participants were achieving discharge-readiness criteria.
Measure: Median (Inter-Quartile Range); unit: score on a scale from 0 to 10
Arm/Group | Normal Saline | Acetaminophen
Number analyzed (Participants) | 31 | 34
score on a scale from 0 to 10
  15 minutes | 9 [7 to 10] | 7 [5 to 9]
  30 minutes: number analyzed (Participants) | 31 | 32
  30 minutes | 8 [6 to 10] | 7 [6 to 8]
  45 minutes: number analyzed (Participants) | 30 | 32
  45 minutes | 7 [5 to 8] | 6 [4 to 8]
  60 minutes: number analyzed (Participants) | 28 | 29
  60 minutes | 5 [3 to 7] | 4 [2 to 6]
  75 minutes: number analyzed (Participants) | 21 | 18
  75 minutes | 5 [4 to 7] | 4 [3 to 6]
  90 minutes: number analyzed (Participants) | 16 | 13
  90 minutes | 5 [3 to 6] | 3 [3 to 6]
  105 minutes: number analyzed (Participants) | 10 | 7
  105 minutes | 5 [3 to 7] | 3 [2 to 8]
  120 minutes: number analyzed (Participants) | 6 | 3
  120 minutes | 6.5 [5 to 7] | 3 [2 to 7]

3. Secondary Outcome: Plasma Stress Markers
Description: Concentration of the plasma stress markers including epinephrine, norepinephrine, cortisol, interleukins (IL) 6, 8 and 10.
Time Frame: Before administration of any drug (after placement of intravenous (IV) line), before surgical incision (in operating room (OR)), and 1 h after arrival in post-anesthesia care unit (PACU)
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Normal Saline | Acetaminophen
Number analyzed (Participants) | 31 | 34
pg/ml
  Epinephrine After IV | 48 [34 to 91] | 65 [42 to 87]
  Epinephrine In OR | 42 [24 to 52] | 58 [37 to 108]
  Epinephrine 1h in PACU | 152 [81 to 255] | 128 [82 to 184]
  Norepinephrine After IV | 643 [546 to 928] | 644 [402 to 900]
  Norepinephrine In OR | 532 [350 to 665] | 547 [341 to 872]
  Norepinephrine 1h in PACU | 689 [444 to 1054] | 884 [533 to 1121]
  Cortisol After IV | 50.5 [30.2 to 76.8] | 54.6 [29.9 to 75.8]
  Cortisol in OR | 45.6 [28.5 to 74.4] | 49 [27.6 to 82.5]
  Cortisol 1h in PACU | 175.9 [90.7 to 212] | 150.1 [84.2 to 212]
  IL-6 after IV | 1.4 [0.9 to 2.4] | 2.3 [1.4 to 3]
  IL-6 in OR | 1.6 [1 to 2.6] | 2 [1.2 to 2.8]
  IL-6 1h in PACU | 7.9 [4.6 to 11.1] | 9.9 [5.6 to 13]
  IL-8 after IV | 8.7 [6.7 to 10.4] | 8.3 [5.7 to 10.7]
  IL-8 in OR | 6.6 [5.5 to 10.1] | 6.4 [4.7 to 8.4]
  IL-8 1h in PACU | 13.7 [9.1 to 23.3] | 12.5 [7.5 to 24]
  IL-10 after IV | 0.6 [0.3 to 1.3] | 1 [0.6 to 1.5]
  IL-10 in OR | 0.5 [0.4 to 1.1] | 1.9 [0.8 to 3.4]
  IL-10 1h in PACU | 1.9 [0.8 to 3.4] | 1.9 [1.3 to 3.3]

4. Secondary Outcome: The Level of C-reactive Protein
Description: Concentration of the plasma C-reactive protein (CRP)
Time Frame: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: pg/ml *1000
Arm/Group | Normal Saline | Acetaminophen
Number analyzed (Participants) | 31 | 34
pg/ml *1000
  CRP after IV | 1062.6 [510.1 to 3741.4] | 1710.9 [714.2 to 3536]
  CRP in OR | 893.4 [370.3 to 2336.4] | 1410.7 [662.8 to 2943.2]
  CRP 1h in PACU | 746.6 [309 to 3861] | 1090.1 [449.2 to 3461.5]

5. Secondary Outcome: Time to Rescue Pain Medication
Description: Time to the first dose of pain medication
Time Frame: From arrival in PACU to the first dose of pain medication is given during 2 hours or until achieving discharge-readiness, whatever comes first, an average of 1 hour.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Normal Saline | Acetaminophen
Number analyzed (Participants) | 31 | 34
minutes | 19 [15 to 28] | 23 [17 to 30]

6. Secondary Outcome: Total Dosage of Post Operative Opioids
Description: Total dosage of post operative opioids (hydromorphone)
Time Frame: From arrival in PACU for 2 hours or until achieving discharge-readiness, whatever comes first, an average of 1 hour.
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | Normal Saline | Acetaminophen
Number analyzed (Participants) | 31 | 34
mg | 1.2 [1 to 1.6] | 1 [0.6 to 1.6]

7. Secondary Outcome: Patient Satisfaction Survey
Description: Survey asking patients about their satisfaction with the experience, pain control, and anesthetic rated on a 5 point Likert scale, with 1 being dissatisfied/unlikely and 5 being most satisfied/very likely. Subscales were summed to receive total score.
Time Frame: For patients going home the day of surgery the survey is given prior to departing the hospital (approx 5 hours post surgery). For those being admitted, the survey is given once discharge criteria are met in the PACU (approx 3 hours post surgery).
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Normal Saline | Acetaminophen
Number analyzed (Participants) | 31 | 34
score on a scale | 4 [3 to 4] | 4 [3 to 4]

8. Secondary Outcome: Number of Participants With Post Operative Nausea and Vomiting
Description: Number of Participants with Post Operative Nausea and Vomiting
Time Frame: From arrival in PACU for 2 hours or until achieving discharge-readiness, whatever comes first, an average of 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Saline | Acetaminophen
Number analyzed (Participants) | 31 | 34
Participants | 9 | 10

9. Secondary Outcome: Number of Participants Requiring Additional Anti-emetics
Description: Number of Participants Requiring Additional Anti-emetics (anti-vomiting)
Time Frame: From arrival in PACU for 2 hours or until achieving discharge-readiness, whatever comes first, an average of 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Saline | Acetaminophen
Number analyzed (Participants) | 31 | 34
Participants | 8 | 7

ADVERSE EVENTS:
Time Frame: From the time patient sign Informed Consent Form for 24 hours or until discharge from the hospital, whatever comes first, an average of 12 hours
Arm/Group | Normal Saline | Acetaminophen
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/47
Other Adverse Events (participants affected / at risk) | 0/41 | 2/47
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Normal Saline (N=41) | Acetaminophen (N=47)
Surgical complication (Surgical and medical procedures) | 0 (0) | 2 (2) — Surgical complication not related to study medication

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-11-11): https://cdn.clinicaltrials.gov/large-docs/87/NCT02832687/Prot_SAP_001.pdf
  • Informed Consent Form (2019-10-09): https://cdn.clinicaltrials.gov/large-docs/87/NCT02832687/ICF_000.pdf